CLINICAL TRIAL: NCT04891406
Title: A Randomised, Cross-over, Relative Bioavailability Study of Nicotine Delivery and Nicotine Extraction From Oral Products (Traditional Snus, Conventional Cigarette and Three Oral Tobacco-free Nicotine Delivery Products)
Brief Title: A Randomised, Cross-over, Relative Bioavailability Study of Nicotine Delivery and Nicotine Extraction From Oral Products
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial Brands PLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: IB-OND-PKZX-01
Record Dates: First submitted 2021-05-12; First posted 2021-05-18 (Actual); Results first posted 2023-10-13 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Fumigant 93; HTR3D protein, human

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- ABCDE (Other): Subjects use product A (ZoneX #2, white tobacco-free nicotine pouch, 5.8 mg nicotine/pouch) for 20 minutes on Day 1, then switch to use product B (ZoneX #3, white tobacco-free nicotine pouch, 10.1 mg nicotine/pouch) for 20 min on Day 2, then product C (Skruf snus fresh slim white, 10.9 mg nicotine/pouch) for 20 min on Day 3, then D (nicotine pouch, 10.6 mg/pouch) on Day 4 and finally E (Marlboro Gold, conventional cigarette, 0.8 mg nicotine/cigarette), smoked in approximately 5 minutes with puffs taken at regular intervals approximately 30 seconds apart, on Day 5.
  Subjects can use their assigned product ad libitum on each study day, after all study assessments are performed, until 10pm. A washout period of product abstinence is observed between products, overnight.
  Interventions: Other: A; Other: B; Other: C; Other: D; Other: E
- BCDEA (Other): Same as previous arm but in a different randomization order.
  Interventions: Other: A; Other: B; Other: C; Other: D; Other: E
- CDEAB (Other): Same as previous arm but in a different randomization order.
  Interventions: Other: A; Other: B; Other: C; Other: D; Other: E
- DEABC (Other): Same as previous arm but in a different randomization order.
  Interventions: Other: A; Other: B; Other: C; Other: D; Other: E
- EABCD (Other): Same as previous arm but in a different randomization order.
  Interventions: Other: A; Other: B; Other: C; Other: D; Other: E

INTERVENTIONS:
Other: A — Use of product A (ZoneX #2, white tobacco-free nicotine pouch, 5.8 mg nicotine/pouch) for 20 minutes
  Other Names: Product A
Other: B — Use of product B (ZoneX #3, white tobacco-free nicotine pouch, 10.1 mg nicotine/pouch) for 20 minutes
  Other Names: Product B
Other: C — Use of product C (Skruf snus fresh slim white, 10.9 mg nicotine/pouch) for 20 minutes
  Other Names: Product C
Other: D — Use of product D (Nicotine pouch, 10.6 mg/pouch) for 20 minutes
  Other Names: Product D
Other: E — Use of product E (Marlboro Gold, conventional cigarette, 0.8 mg nicotine/cigarette) for approximately 5 minutes
  Other Names: Product E

SUMMARY:
This study is a randomised cross-over, open-label, confinement study conducted in 24 male or female snus and cigarette consumers. The study investigates 5 different nicotine containing products in a cross-over fashion. The study incorporates pharmacokinetics evaluation, nicotine extraction evaluation, subjective questionnaire assessments as well as safety evaluation.

During the study participation, subjects come for two visits to the clinic, including a 5-day confinement period.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) ≥ 18.0 and ≤ 30.0 kg/m
* Clinically normal medical history, physical findings, vital signs, ECG and laboratory values at the time of screening, as judged by the Investigator
* Dual user of snus and conventional cigarettes for ≥1 year, with a minimum weekly consumption of two or more snus cans and >5 cigarettes, and who is willing and able to use brands with nicotine content ≥1%

Exclusion Criteria:

* History of any clinically significant disease or disorder
* Any clinically significant illness, medical/surgical procedure or trauma within 4 weeks of the first use of IP
* Positive for HIV, hepatitis B or C
* After 10 minutes supine rest at the time of screening, any vital signs values outside the following ranges:

  * Systolic blood pressure <90 or >140 mmHg, or
  * Diastolic blood pressure <50 or >90 mmHg, or
  * Pulse <40 or >90 bpm
* Alcohol or drug abuse
* Use, or history of use of anabolic steroids
* Allergy/hypersensitivity to drugs with a similar chemical structure or class to nicotine
* Excessive caffeine consumption (daily intake of >5 cups)
* Female subjects who are pregnant or breastfeeding

Ages: 19 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-01-20 (Actual); Study Completion 2021-01-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- CTC Clinical Trial Consultants AB (CTC), Uppsala, Sweden

REFERENCES:
- [Derived] Chapman F, McDermott S, Rudd K, Taverner V, Stevenson M, Chaudhary N, Reichmann K, Thompson J, Nahde T, O'Connell G. A randomised, open-label, cross-over clinical study to evaluate the pharmacokinetic, pharmacodynamic and safety and tolerability profiles of tobacco-free oral nicotine pouches relative to cigarettes. Psychopharmacology (Berl). 2022 Sep;239(9):2931-2943. doi: 10.1007/s00213-022-06178-6. Epub 2022 Jun 23. PMID 35732751

RESULTS

PARTICIPANT FLOW:
Groups:
- ABCDE: Subjects use product A (ZoneX #2, white tobacco-free nicotine pouch, 5.8 mg nicotine/pouch) for 20 minutes on Day 1, then switch to use product B (ZoneX #3, white tobacco-free nicotine pouch, 10.1 mg nicotine/pouch) for 20 min on Day 2, then product C (Skruf snus fresh slim white, 10.9 mg nicotine/pouch) for 20 min on Day 3, then D (nicotine pouch, 10.6 mg/pouch) on Day 4 and finally E (Marlboro Gold, conventional cigarette, 0.8 mg nicotine/cigarette), smoked in approximately 5 minutes with puffs taken at regular intervals approximately 30 seconds apart, on Day 5.
  Subjects can use their assigned product ad libitum on each study day, after all study assessments are performed, until 10pm. A washout period of product abstinence is observed between products, overnight.
  A: Use of product A (ZoneX #2, white tobacco-free nicotine pouch, 5.8 mg nicotine/pouch) for 20 minutes
  B: Use of product B (ZoneX #3, white tobacco-free nicotine pouch, 10.1 mg nicotine/pouch) for 20 minutes
  C: Use of product C (Skruf snus fresh slim white, 10.9 mg nicotine/pouch) for 20 minutes
  D: Use of product D (Nicotine pouch, 10.6 mg/pouch) for 20 minutes
  E: Use of product E (Marlboro Gold, conventional cigarette, 0.8 mg nicotine/cigarette) for approximately 5 minutes
Period: Overall Study
Arm/Group | ABCDE | BCDEA | CDEAB | DEABC | EABCD
Started | 5 | 5 | 5 | 5 | 4
Completed | 5 | 4 | 5 | 5 | 3
Not Completed | 0 | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ABCDE | BCDEA | CDEAB | DEABC | EABCD | Total
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 4 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.2 (4.3) | 25.0 (1.4) | 32.6 (10.8) | 34.2 (10.0) | 38.5 (14.2) | 30.4 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 1 | 2 | 3
  Male | 5 | 5 | 5 | 4 | 2 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1 | 0 | 2
  Not Hispanic or Latino | 5 | 4 | 5 | 4 | 4 | 22
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 25.7 (4.4) | 21.2 (2.1) | 24.6 (3.6) | 24.5 (2.1) | 25.1 (4.8) | 24.2 (3.6)

OUTCOME MEASURES:

1. Primary Outcome: Nicotine Cmax
Description: Maximum plasma concentration of nicotine (Cmax)
Time Frame: Pre-use and at 2, 5, 7, 15, 20, 30, 45, 60, 90 minutes, and 2, 4, 6 and 8 hours post use start
Population: The analysis population represents all subjects who used a specific product. The overall number of participants analyzed for each product is therefore different from the number of participants in each arm provided in the Participant Flow module.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Product A: Subjects who used product A (ZoneX #2, white tobacco-free nicotine pouch, 5.8 mg nicotine/pouch) for 20 minutes
- Product B: Subjects who used product B (ZoneX #3, white tobacco-free nicotine pouch, 10.1 mg nicotine/pouch) for 20 min
- Product C: Subjects who used product C (Skruf snus fresh slim white, 10.9 mg nicotine/pouch) for 20 min
- Product D: Subjects who used Product D (nicotine pouch, 10.6 mg/pouch) for 20 min
- Product E: Subjects who used Product E (Marlboro Gold, conventional cigarette, 0.8 mg nicotine/cigarette), smoked in approximately 5 minutes
Arm/Group | Product A | Product B | Product C | Product D | Product E
Number analyzed (Participants) | 21 | 22 | 22 | 23 | 22
ng/mL | 5.154 (1.662) | 7.856 (2.451) | 9.553 (4.083) | 12.51 (4.377) | 11.60 (5.171)

2. Primary Outcome: Nicotine AUCt
Description: Area under the plasma nicotine concentration-time curve at the last timepoint measured (AUCt)
Time Frame: Pre-use and at 2, 5, 7, 15, 20, 30, 45, 60, 90 minutes, and 2, 4, 6 and 8 hours post use start
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Product A | Product B | Product C | Product D | Product E
Number analyzed (Participants) | 21 | 22 | 22 | 23 | 22
h*ng/mL | 12.23 (4.996) | 18.35 (8.180) | 21.13 (11.38) | 31.31 (13.98) | 19.60 (10.75)

3. Secondary Outcome: Nicotine Extraction
Description: Extraction fraction (%) of nicotine in used product pouches after 20 minutes of use.
Time Frame: 20 minutes
Population: The analysis population represents all subjects who used a specific product. The overall number of participants analyzed for each product is therefore different from the number of participants in each arm provided in the Participant Flow module.
  Only analyzed for pouch products (A, B, C and D), not for Product E (conventional cigarette).
Measure: Mean (Standard Deviation); unit: Percent of nicotine used
Arm/Group | Product A | Product B | Product C | Product D
Number analyzed (Participants) | 22 | 22 | 22 | 23
Percent of nicotine used | 13.47 (5.321) | 14.31 (8.181) | 12.56 (5.010) | 18.61 (8.608)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the start of the first Investigational Product use until the end-of-study visit (7 Days).
Description: The number of participants at risk represents all subjects who used a specific product. The overall number of participants analyzed for each product is therefore different from the number of participants in each arm provided in the Participant Flow module.
Arm/Group | Product A | Product B | Product C | Product D | Product E
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/23 | 0/22 | 0/23 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/23 | 0/22 | 0/23 | 0/22
Other Adverse Events (participants affected / at risk) | 3/22 | 0/23 | 1/22 | 1/23 | 3/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Product A (N=22) | Product B (N=23) | Product C (N=22) | Product D (N=23) | Product E (N=22)
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Thrombophlebitis (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-08-26): https://cdn.clinicaltrials.gov/large-docs/06/NCT04891406/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-02): https://cdn.clinicaltrials.gov/large-docs/06/NCT04891406/SAP_001.pdf